CLINICAL TRIAL: NCT05482464
Title: Effect of Daily Consumption of Glycomacropeptide on Gut Microbiome and Blood Functional Proteome of Subjects With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: BUILD Dairy (Unknown); Agropur (Unknown)
Responsible Party: Principal Investigator, Dave Dallas, Assistant Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2021-1186
Record Dates: First submitted 2022-04-06; First posted 2022-08-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Casein glycomacropeptide (CGMP) (Other): The subjects will receive a daily oral intake of CGMP-protein-shake for 3 weeks with a 1 week wash-in and a 3 week wash-out.
  Intervention: Dietary Supplement: Casein glycomacropeptide (CGMP)
  Interventions: Dietary Supplement: Casein glycomacropeptide (CGMP)

INTERVENTIONS:
Dietary Supplement: Casein glycomacropeptide (CGMP) — Casein glycomacropeptide (CGMP) supplementation for 3 weeks

SUMMARY:
This study investigates the use of glycomacropeptide (GMP) as a means to manipulate the gut microbiome, metabolome and protein profile of subjects with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
In vitro assays show that GMP strongly promotes the growth of beneficial bacteria including Bifidobacterium breve, B. bifidum, B. infantis and Lactococcus lactis. GMP also binds to pathogenic bacteria and prevents their adhesion to intestinal cells, which could prevent enteric infection. GMP also modulates the inflammatory response of key gut immune cells called macrophages. However, the extent to which daily consumption of GMP alters the gut microbiome, metabolome and protein profile of subjects with IBS remains unknown.

This study will investigate how daily GMP consumption can alter the gut microbiome, metabolome and protein profile of subjects with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* IBS diagnosis with Rome IV criteria
* People who have a primary care provider

Exclusion Criteria:

* Lactose or milk protein intolerance
* Any known other gastrointestinal disease or disorder beyond IBS, or major gastrointestinal surgery
* Habitual use of laxatives or antacids
* Pregnant or nursing.
* Use of pre or probiotics within one month prior to the study
* Use of antibiotics within one month prior to the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Measure the inflammatory markers in stool and blood using immunology multiplex assay | Baseline, GMP feeding week 1, 2 and 3 and post study without GMP feeding week 1, 2 and 3
  Change in levels of inflammatory markers (GM-CSF, IFN-γ, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17A, IL-17F, IL-17E/IL-25, IL-21, IL-22, IL-23, IL-27, IL-28A, IL-31, IL-33, MIP-3α/CCL20, TNF-α and TNFβ) in stool and blood using immunology multiplex assay
Stool sample based gut microbiome composition using 16S rRNA gene sequencing | Baseline, GMP feeding week 1, 2 and 3 and post study without GMP feeding week 1, 2 and 3
  Change in stool sample based gut microbiome composition using 16S rRNA gene sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Milam Hall, Room 001, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No